CLINICAL TRIAL: NCT07188792
Title: The Effect of Horticultural Therapy Applied to Caregivers of Hemodialysis Patients on Perceived Stress, Well-Being Level, and Care Burden: A Randomized Controlled Trial
Brief Title: The Effect of Horticultural Therapy on Stress, Well-Being, and Care Burden in Hemodialysis Caregivers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mahmut Coban, lecturer, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/210 -63
Record Dates: First submitted 2025-09-08; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Hemodialysis Patients
Keywords: perceived stress; caring; maintenance burden; hemodialysis patient; horticultural therapy
MeSH Terms: interventions — Horticultural Therapy

STUDY DESIGN:
Intervention Model Description: The study population consisted of 120 caregivers receiving treatment in the hemodialysis unit at Bingöl State Hospital; the sample consisted of 82 caregivers who met the study criteria and agreed to participate in the study. The sample size for the study was calculated as 70 using the G*Power 3.1 program, taking into account similar studies, a 5% effect size, 95% reliability, and 80% theoretical power. To prevent participants from withdrawing from the study at any stage, 12 more individuals (15% more than the sample size) were added to the predetermined sample, resulting in a total of 82 participants. Those who agreed to participate after obtaining verbal consent from these individuals were included in the sample. The caregiver assignment to the experimental or control groups was determined at the beginning of the study using the Random Allocation Software 1.0.0 package program.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Single blindness is achieved by not specifying which section is specified during the data collection process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): The Caregiver Identification Form, Perceived Stress Scale, General Well-Being Scale and Zarit Caregiver Burden Scale were applied to the experimental and control groups. In the study, horticultural activities prepared with literature support and expert opinions as a nursing intervention were applied to the experimental group once a week for 12 weeks.
  Interventions: Other: HORTICULTURAL THERAPY
- CONTROL GROUP (No Intervention): No ınterventıon was made to the control group durıng the study. After the gardening care activity in which the experimental system was applied, the Perceived Stress Scale, General Well-Being Scale and Zarit Caregiving Burden Scale were administered to the individuals in the experimental and control groups in order to measure the post-test data.

INTERVENTIONS:
Other: HORTICULTURAL THERAPY — * Introduction
  * Explanation of the training content for horticultural activities using visual materials
  * Explanation of the program's scope, duration, and expected participant roles and responsibilities
  Arms: EXPERIMENTAL GROUP

SUMMARY:
This research is a randomized controlled single-blind experimental study aiming to evaluate the effect of horticultural therapy on stress, well-being, and caregiver burden among caregivers of hemodialysis patients. The study will be conducted between April-July 2025 with caregivers of patients receiving hemodialysis treatment at Bingöl State Hospital. The sample of the study will consist of 82 caregivers, randomly assigned into experimental and control groups. After obtaining verbal and written consents from all participants, the Introductory Information Form, Perceived Stress Scale, General Well-Being Scale, and Zarit Burden Interview will be applied as pre-test. The experimental group will participate in horticultural therapy activities once a week for 12 weeks, while no intervention will be given to the control group during this period. Following the intervention, post-test measurements will be administered to both groups using the same instruments. In addition, feedback will be collected from caregivers in the experimental group regarding the research process. After the study is completed, the same intervention will also be offered to the control group to ensure ethical responsibility. Data obtained will be analyzed using SPSS 22.00 package program. Ethical principles will be observed throughout the study, ethics committee approval has been obtained, and the Helsinki Declaration of Human Rights will be adhered to. The results are planned to be presented at an international congress and published in an SCI/SSCI-indexed journal, contributing to the scientific literature.

DETAILED DESCRIPTION:
INTRODUCTION Chronic kidney failure (CKD) is an important health problem worldwide, with a rising prevalence particularly in low- and middle-income countries. The number of patients with kidney failure doubles approximately every seven years. According to World Health Organization data, nearly 850 million people globally are affected by kidney disease, creating a significant health burden and economic cost. In Türkiye, the prevalence of chronic kidney disease is estimated to be around 15%.

One of the most commonly used treatment methods in patients with chronic kidney failure is dialysis, defined as the removal of excess fluids and waste products in situations where the kidneys are unable to perform their functions due to dysfunction. It is estimated that approximately 2-3 million people worldwide are receiving hemodialysis/dialysis treatment. In the United States, about 700,000 end-stage kidney failure patients exist, of whom 65% are treated with hemodialysis. In Japan, as of the end of 2018, 339,841 hemodialysis patients were reported. In Türkiye, according to 2022 data, more than 120,000 patients were receiving hemodialysis treatment, and records show that there are more than 500 dialysis centers nationwide.

The lives of caregivers of individuals undergoing hemodialysis treatment are negatively affected in many aspects. Caregivers frequently experience problems such as fatigue, pain, weakness, sleep disorders, depression, anxiety, burnout, social life restrictions, and economic difficulties. In addition, studies have reported that caregivers show decreased engagement in preventive health behaviors, face increased health problems, and are at higher risk of mortality.

For centuries, the healing power of nature has been emphasized, and it is well known that natural environments reduce stress in patients. Horticultural therapy encompasses a multidimensional process. Individuals not only spend time in green spaces but also actively interact with plants, engage in psychotherapeutic experiences, and improve their decision-making processes. Planting seeds, witnessing them blossom, and observing the growth of plants and trees inspire people with hope for life. It is believed that nature and humans are inseparable parts of life, and therefore, nature creates a positive impact on individuals.

Furthermore, horticultural therapy, which involves green spaces and plants, has been reported as an important rehabilitation method in the relationship between nature and the promotion of general well-being. The program carried out in this study aims to reduce stress and mental fatigue; to enhance self-esteem and self-efficacy; to contribute to well-being; and to alleviate caregiver burden.

Keywords: Perceived stress, caregiver, care burden, hemodialysis patient, nursing, horticultural therapy, well-being.

Research Hypotheses:

H1: Horticultural therapy applied to caregivers of hemodialysis patients reduces caregivers' stress levels.

H2: Horticultural therapy applied to caregivers of hemodialysis patients increases caregivers' well-being levels.

H3: Horticultural therapy applied to caregivers of hemodialysis patients reduces caregiver burden.

MATERIALS AND METHODS

Type of Research:

This study is a randomized controlled, single-blind, pretest-posttest, control group experimental research aimed at evaluating the effects of horticultural therapy on the perceived stress, well-being, and caregiver burden of caregivers of hemodialysis patients.

Research Location and Time:

The study was conducted between April 20, 2025, and July 20, 2025, with caregivers of patients receiving hemodialysis treatment at Bingöl State Hospital, in an area designated by the hospital.

The garden area, approximately 300 m², is located on the east side of the hospital building and is a semi-open space integrated with the natural environment. It consists of three sections with concrete-paved walkways and a balanced distribution of green vegetation. Normally not open to public use, this area was reserved exclusively for the experimental group during the research period and opened to all caregivers after the study was completed. To ensure safety and privacy, the area was surrounded by security tape. Various seating arrangements (benches and shaded areas) were provided to allow caregivers opportunities for rest and social interaction.

The landscaping was designed to contribute to the psychosocial relaxation of users. The area was regularly maintained in accordance with cleaning standards throughout the study period. In addition, by providing a safe, calm, and peaceful environment, the research process progressed smoothly.

Population and Sample:

The study population consisted of 120 caregivers of patients receiving treatment at the Hemodialysis Unit of Bingöl State Hospital. The study sample consisted of 82 caregivers who met the inclusion criteria and agreed to participate in the study.

Based on similar studies, the sample size was calculated as 70 using the G*Power 3.1 program with a 5% effect size, 95% confidence, and 80% power. To prevent attrition, 12 more participants (15% more than the calculated size) were added, resulting in a total of 82 caregivers. Participants who gave verbal consent were included in the study.

The assignment of caregivers to experimental and control groups was carried out at the beginning of the study using the Random Allocation Software 1.0.0. A total of 82 caregivers were randomly assigned to experimental and control groups with the computer-based Research Randomizer program. Group assignments were made by an independent observer, and in line with the single-blind principle, caregivers were not informed of their group allocation. Written and verbal consent was obtained, and pretests were administered afterward. Analyses showed no significant differences between the groups, confirming homogeneity.

Inclusion Criteria:

Being the primary caregiver of a patient receiving treatment in the hemodialysis unit, Having provided active care for at least six months, Not having a physical condition preventing participation in horticultural activities, Not having a psychiatric disorder, Being able to communicate and collaborate, Regularly attending at least 80% of the horticultural activity sessions (nine sessions).

Exclusion Criteria:

Having a physical illness preventing participation in gardening activities, Having a psychiatric disorder, Being at risk of transfer with their patient to another dialysis center during the study period, Lack of continuity in caregiving.

Study Variables:

Dependent Variables: Mean scores of the Perceived Stress Scale, General Well-Being Scale, and Zarit Caregiver Burden Scale.

Independent Variable: Horticultural therapy activities. Control Variables: Age, gender, marital status, education level, caregiving duration.

Data Collection Tools:

Caregiver Introduction Form: A 16-item form prepared based on the literature. Perceived Stress Scale: 10 items, Likert scale 1-5. Higher scores = higher stress.

General Well-Being Scale : 13 items, 5-point Likert. Higher scores = higher well-being.

Zarit Caregiver Burden Scale: 22 items, Likert scale 1-5. Higher scores = higher caregiver burden.

Nursing Interventions:

Horticultural activities were designed with reference to the literature and expert opinions, and implemented as a nursing intervention once a week for 12 weeks in the experimental group. No intervention was applied to the control group.

The flowers used in the study (Tagates Erecta, Celosia Cristata, Petunia Grandiflora) were selected for their adaptability to the regional climate, low water requirements, variety of colors, and ability to grow in different soil types.

Activities were carried out with caregivers accompanying patients during dialysis sessions. Monday and Tuesday were designated as intervention days. Caregivers in the experimental group participated once a week for 12 weeks. The first session was held in the hospital training room, while the remaining sessions were held in the designated hospital garden area. Each session lasted 90 minutes (30 minutes of activity + 30 minutes break + 30 minutes of activity).

The activities were conducted by the researcher, who had completed the training program "Horticultural Therapy Approach Based on Human-Health-Nature" held at Ordu University (February 5-9, 2024) under the TÜBİTAK 2237/A Scientific Education Activities Support Program.

Data Collection:

Pretest: Conducted between April 15-20, 2025. The Caregiver Introduction Form, Perceived Stress Scale, General Well-Being Scale, and Zarit Caregiver Burden Scale were administered face-to-face. Average duration: 25 minutes.

Posttest: Conducted between July 20-25, 2025. The same scales were administered face-to-face. Average duration: 25 minutes. Group allocation was not disclosed to participants, ensuring single-blindness.

ELIGIBILITY:
Inclusion Criteria:

* Being the primary caregiver for a patient receiving treatment in a hemodialysis unit,
* Having provided active care for at least six months,
* Not having a physical condition that would prevent participation in horticultural activities,
* Not having a psychiatric illness,
* Being able to communicate and be open to collaboration,
* Having regularly attended at least 80% (nine) of the horticultural activity sessions.

Exclusion Criteria:

* Those with a physical illness that would prevent them from participating in gardening-based activities,
* Those with a psychiatric illness,
* Those whose caregiver may be transferred to another dialysis center along with their patient during the study period,
* Caregivers with no continuity of care.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Caregiver Introduction Form | baseline
  This form was prepared by researchers based on literature. It consists of 16 questions covering the sociodemographic characteristics of caregivers (age, gender, family type, marital status, number of children, number of family members, occupation, economic status, education level, place of residence, number of years the patient has been receiving dialysis treatment, degree of closeness to the caregiver, length of caregiving, duration of daily caregiving, other caregivers in the family, and presence or absence of chronic illness).

SECONDARY OUTCOMES:
Perceived Stress Scale | at the beginning and at the end of the 12-week study
  The scale, developed by Cohen et al. (1983) and adapted into Turkish by Erci (2006), aims to determine perceived stress. The scale consists of 10 items, each scored from 1 to 5: never (1), almost never (2), sometimes (3), often (4), and very often (5). Four items are scored positively, and six items are scored negatively, with total scores ranging from 10 to 50. Higher scores indicate higher levels of stress. The Cronbach's alpha for the adapted version of the scale is 0.88.

OTHER OUTCOMES:
General Well-Being Scale | at baseline and at the end of the 12-week study
  Developed by Longo et al. (2018) and adapted into Turkish by Kalafatoğlu and Çelik (2020), the scale measures general well-being. The items are designed on a 5-point Likert-type scale ranging from "Not at all applicable" to "Completely applicable." It is a single-factor, 13-item, five-point Likert-type scale (1 - Completely Disagree - 5 - Completely Agree). The lowest possible score is 5, and the highest is 65. The scale's Cronbach's alpha is 0.90. It has been reported that higher scores indicate higher levels of general well-being.
Zarit Caregiving Burden Scale | at baseline and at the end of the 12-week study
  The Zarit Caregiver Burden Scale, developed by Zarit et al. (1980), was adapted into Turkish by İnci and Erdem (2008). It is used to identify the problems experienced by caregivers of individuals in need of care. The scale consists of 22 questions measuring the impact of caregiving on a person's life. It uses a Likert-type scale ranging from 1 to 5, with scores ranging from never, rarely, sometimes, often, or almost always. The lowest possible score is 0, and the highest is 88. Higher scores indicate an increased caregiver burden. The Cronbach's alpha value for the scale, which is considered more appropriate for a single-dimensional approach, was found to be 0.95.

CONTACTS AND LOCATIONS:
Overall Officials: DİLEK KILIÇ, Principal Investigator — Ataturk University; GÜLNAZ ATA, Principal Investigator — TOKAT GAZİOSMANPAŞA UNIVERSITY
Locations (1):
- Atatürk Üniverty, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No